CLINICAL TRIAL: NCT05891379
Title: Effectiveness and Safety of Inebilizumab in the Acute Phase of Neuromyelitis Optica Spectrum Disorders-a Multicentric, Prospective, Real Word Study
Brief Title: Inebilizumab in Acute Neuromyelitis Optica Spectrum Disorders
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: XMEC-2023-003
Record Dates: First submitted 2023-05-24; First posted 2023-06-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica Spectrum Disorder; inebilizumab; observational study
MeSH Terms: conditions — Neuromyelitis Optica | interventions — inebilizumab; Immunosuppressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected before the treatment and at the last visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed group: intravenous Intravenous methylprednisolone (IVMP) plus intravenous inebilizumab
  Interventions: Drug: Inebilizumab
- Non-exposed group: IVMP plus oral immunosuppressant (Mycophenolate Mofetil or Azathioprine)
  Interventions: Drug: oral immunosuppressant

INTERVENTIONS:
Drug: Inebilizumab — Inebilizumab: 300mg IV on Day1 and Day 15. The first dose of inelizumab is given during IVMP.
  Groups: Exposed group
Drug: oral immunosuppressant — Oral immunosuppressants (azathioprine or mycolate mofetil) are initiated during IVMP.
  Groups: Non-exposed group

SUMMARY:
This study is aimed to observe the effectiveness and safety of inebilizumab in the acute phase of neuromyelitis optica spectrum disorders.

DETAILED DESCRIPTION:
This is a a multicentric, prospective, real word study of inebilizumab in NMOSD acute attack compared with oral immunosuppressant. A total of 50 patients will be enrolled at approximately 10 centers around China.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years with anti-AQP4-IgG seropositive NMOSD as defined by 2015 NMOSD diagnostic criteria by IPND (International Panel for NMO Diagnosis); 2. In the acute phase of NMOSD (definition of acute phase: new neurological symptoms or aggravation of existing symptoms within 30 days before screening, lasting at least 24 hours without with fever); 3. Patients who plan to receive or are receiving intravenous methylprednisolone therapy; 4. Expanded disability status scale (EDSS) score ≤ 8 and ≥ 2.5 during the screening period; 5. Able and willing to give written informed consent; 6. Women of childbearing potential who agree to use adequate contraception during the study.

Exclusion Criteria:

* 1. Lactating and pregnant females; 2. Participate in other interventional studies within 30 days before screening or within 5 half-lives of the investigational agent before enrollment; 3. Combined with severe mental disorders and other conditions and unable to cooperate with follow-up; 4. History of malignancies; 5. Received plasma exchange, immunoadsorption or intravenous immunoglobulin therapy within 1 month before screening; 6. Patients with negative hepatitis B surface antibody (HBsAg) and positive hepatitis B core antibody (HBcAb), or HBsAg-positive virus carriers, or patients with active tuberculosis or positive tuberculosis screening without appropriate treatment history; 7. Other situations that researchers think are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NMOSD patients with acute attacks
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score from baseline | 6 months
  Change in Expanded Disability Status Scale (EDSS) score from baseline at the last visit(EDSS : Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score from baseline | 1 months, 3 months
  Change in Expanded Disability Status Scale (EDSS) score from baseline at month 1, month 3(EDSS : Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).
Percentage of Participants With Disability Improvement | 6 months
  Disability improvement is defined as a reduction in EDSS score of: A) >=1.0 from the baseline EDSS score when the baseline score was <=5.5 B) >= 0.5 when the baseline EDSS score > 5.5(EDSS : Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).
Change in modified Rankin score (mRS) from baseline | 1 months, 3 months, 6 months
  Change in modified Rankin score (mRS) from baseline at month 1, month 3, month 6(mRS : Minimum Score 0, Maximum score 6, higher scores mean a worse outcome).
Time to first relapse | 6 months
Number of New, and/or Enlarging T2 Hyperintense Lesions Detected by Magnetic Resonance Imaging (MRI) | 6 months
  Number of New, and/or Enlarging T2 Hyperintense Lesions Detected by Magnetic Resonance Imaging (MRI) at the last visit
Change in Timed 25 Foot Walk Test from baseline | 1 months, 3 months , 6 months
  Change in time taken to complete the timed 25 foot walk test from baseline
Number of NMOSD attacked related rescue treatment | 6 months
Change in serum GFAP levels from baseline | 6 months
  Change in serum GFAP levels from baseline at the last visit
Change in AQP4-ab titers from baseline | 6 months
  Change in AQP4-ab titers from baseline at the last visit
Change in Low-contrast Visual Acuity (LCVA) from baseline | 3 months, 6 months
  Change in Low-contrast Visual Acuity (LCVA) at month 3, month 6)(The LCVA test is used to determine the number of letters that can be read on a standardized low-contrast Landolt C Broken Rings Chart held at a distance of 3 meters).
Changes in EQ-5D-5L scores from baseline | 1 month, 3 months ,6 months
  Changes in EQ-5D scores from baseline at month 1 month, month 3 , month 6(EQ-5D-5L: Minimum Score 5, Maximum score 25, lower scores mean a better quality of life).
Change in retinal nerve fiber layer (RNFL) loss from baseline | 3 months ,6 months
  Change in retinal nerve fiber layer (RNFL) loss measured by optical coherence tomography (OCT) from baseline at month 1, month 3，month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No